CLINICAL TRIAL: NCT07119411
Title: ICU Background Early Awareness for Critical deterioratiON (BEACON)
Brief Title: ICU Background Early Awareness for Critical deterioratiON
Acronym: BEACON
Status: Not yet recruiting | Type: Observational
Sponsor: ETH Zurich (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2025-00623
Record Dates: First submitted 2025-07-16; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Failure; Circulatory Failure; Mortality; Organ Dysfunction; Organ Failure, Multiple
Keywords: icu; respiratory failure; circulatory failure; early warning system; prevention; prediction; risk prediction; organ failure; multi-organ failure; win-ratio; ICU Beacon
MeSH Terms: conditions — Respiratory Insufficiency; Shock; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Patients are admitted to the ICU and received the standard of care without the availability of Beacon
- Study Group: Patients are admitted to the ICU and received the standard of care with the additional availability of Beacon by treating clinicians.
  Interventions: Other: ICU Beacon

INTERVENTIONS:
Other: ICU Beacon — Availability of a proprietary clinician awareness for potential organ deterioration software to treating clinicians (ICU Beacon) in addition to the standard of care.
  Other Names: Beacon
  Groups: Study Group

SUMMARY:
The study will compare ICU sub-units, those with additional support of a clinician awareness system, ICU Beacon, and those receiving the standard of care. The win-ratio composite outcome will be assessed by comparing patients by study group and stratified by APACHE score at admission.

DETAILED DESCRIPTION:
Single-center, stratified, cluster-randomized (the ICU units will be randomized) crossover analysis with outcome-assessor blinding. The analysis will be conducted in the adult intensive care units (ICUs) of Inselspital, Bern, comprising two distinct ICU units: the Blue and the Yellow ICU Unit. Each unit contains two sub-units, which will serve as the clustering units for randomization. The study follows a two-phase design. In the initial phase, sub-units within each ICU unit will be randomly allocated in a 1:1 ratio to either the additional BEACON scoring group or control group. Patients admitted to sub-units allocated to the BEACON group will receive standard care plus BEACON scores, while those admitted to control group will receive standard care only. After predefined cluster periods, allocations will be swapped between the BEACON and control groups. A wash-out period of two weeks will be observed between swaps to minimize carryover effects. During the wash-out period, no new study patients will be enrolled. Once the swap is complete, only newly admitted patients will be enrolled under the sub-unit's new allocation. Patients still occupying sub-units from the preceding period will be censored from the study at the time of the swap and excluded from outcome analysis beyond that point. The same approach will be applied for patients who will be transferred from one unit to a different unit during the ICU admission for logistical/organizational reasons. Importantly, individual patients will only be exposed to one analysis condition-either the BEACON or control-based on the bed allocation at the time of their admission. Only the sub-units themselves undergo crossover, ensuring temporal balance while maintaining patient-level exposure to a single condition.

ELIGIBILITY:
Inclusion Criteria:

* admission to intensive care unit

Exclusion Criteria:

* age < 18 years
* presence of documented refused general consent form (at database closure)
* admission for the sole purpose of dying/organ donation or evaluation of such

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes all patients admitted to the Inselspital Bern ICU, not fulfilling any of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 1962 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to determine whether BEACON improves ICU sub-unit performance, i.e. reduces total mortality and/or mitigates severity of organ failures in an adult university ICU setting. | Patient data up to 28 days post admission will be collected to support analysis.
  Determined by a stratified clustered hierarchical win ratio. Patient data is clustered by ICU sub-unit and stratified by APACHE score. For each stratum, each patient in the study group is compared with all patients in the control group within that same stratum. Levels are assessed up to 28 days after admission. The hierarchical levels are:
  1. All-cause mortality;
  2. Number of organ systems failed (respiratory, cardiovascular, coagulation, liver, renal) with SOFA scores newly increasing to 3 points during the ICU stay; and
  3. Sum of highest circulatory and respiratory SOFA scores during the ICU stay, independently assessed and subsequently summed.
  If one patient "wins" at the first level (i.e., is alive while the other is dead), the comparison is decided. If a tie occurs (both alive or both dead at at 28 days), the next level is compared, and so forth. This approach prioritizes the most clinically serious outcome (mortality), while capturing organ dysfunction at different levels.

SECONDARY OUTCOMES:
Time free of circulatory failure and alive at 28 days | Patient data up to 28 days post admission will be collected to support analysis.
  Described by the total number of days the patient was alive and free of circulatory failure within the first 28 days after admission. Circulatory failure is defined as: lactate >= 2 mmol/L and MAP <= 65 mmHg or receipt of vasopressors/inotropes.
Time free of respiratory failure and alive at 28 days | Patient data up to 28 days post admission will be collected to support analysis.
  Described by the total number of days the patient was alive and free of respiratory failure within the first 28 days after admission. Respiratory failure is defined as: (PaO2/FiO2 ratio < 150 mmHg).
All cause mortality at 28 days | Patient data up to 28 days post admission will be collected to support analysis.
  Mortality from any cause within 28 days following ICU admission.
Mean total SOFA score over ICU stay | Patient data up to 28 days post admission will be collected to support analysis.
  The mean SOFA score including all organ systems through the duration of the ICU admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Inselspital - Universitätsspital Bern, Bern, Switzerland

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT07119411/SAP_000.pdf